CLINICAL TRIAL: NCT05859945
Title: A Critical Analysis of Hepatocellular Carcinoma Trials: Perspectives From Patient Experiences
Brief Title: Navigating the Clinical Trial Process for Hepatocellular Carcinoma
Status: Not yet recruiting | Type: Observational
Sponsor: Power Life Sciences Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 82127001
Record Dates: First submitted 2023-05-05; First posted 2023-05-16 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2023-05

CONDITIONS: Hepatocellular Carcinoma
Keywords: hepatocellular carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Clinical trials can sometimes favor certain demographic groups. Additionally, there is limited research that delves into the factors that influence participation in clinical study, both positive and negative.

The goal is to identify the obstacles and challenges that prevent participation in hepatocellular carcinoma clinical research, as well as the reasons for withdrawal or discontinuation.

Insights gained from this study will ultimately benefit those with hepatocellular carcinoma who may be invited to participate in clinical research in the years to come.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with hepatocellular carcinoma
* Willing to comply with all study related procedures and assessments
* Capable of giving signed informed consent, which includes compliance with requirements and restrictions listed in the informed consent form (ICF) and in the protocol

Exclusion Criteria:

* No documented diagnosis of hepatocellular carcinoma
* Any serious and/or unstable pre-existing medical disorders
* Pregnant or lactating woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with hepatocellular carcinoma who are actively considering participating in an observational clinical study, but have not yet completed enrollment and randomization.
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Rate of patients who decide to enroll in a hepatocellular carcinoma clinical study. | 3 months
Number of hepatocellular carcinoma study participants who remain in clinical trial until completion. | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael B Gill, Study Director — Power Life Sciences Inc.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Frenette C, Gish R. Targeted systemic therapies for hepatocellular carcinoma: clinical perspectives, challenges and implications. World J Gastroenterol. 2012 Feb 14;18(6):498-506. doi: 10.3748/wjg.v18.i6.498. PMID 22363115
- [Background] Haber PK, Puigvehi M, Castet F, Lourdusamy V, Montal R, Tabrizian P, Buckstein M, Kim E, Villanueva A, Schwartz M, Llovet JM. Evidence-Based Management of Hepatocellular Carcinoma: Systematic Review and Meta-analysis of Randomized Controlled Trials (2002-2020). Gastroenterology. 2021 Sep;161(3):879-898. doi: 10.1053/j.gastro.2021.06.008. Epub 2021 Jun 12. PMID 34126063
- [Background] Luo XY, Wu KM, He XX. Advances in drug development for hepatocellular carcinoma: clinical trials and potential therapeutic targets. J Exp Clin Cancer Res. 2021 May 18;40(1):172. doi: 10.1186/s13046-021-01968-w. PMID 34006331

DOCUMENTS (1):
  • Informed Consent Form (2023-05-05): https://cdn.clinicaltrials.gov/large-docs/45/NCT05859945/ICF_000.pdf